CLINICAL TRIAL: NCT01213030
Title: Clinical Evaluation of the New Hypoxia Imaging Agent HX4
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Yi Hui Guan, PET Center, Huashan Hospital, Fudan University, Shanghai, China 200235, Fudan University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HX4-FMISO
Record Dates: First submitted 2009-08-14; First posted 2010-10-01 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer; Lung Cancer; Liver Cancer
Keywords: HX4; [F-18]HX4; FMISO; [F-18]FMISO; Solitary Tumor; Hypoxia
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Liver Neoplasms; Hypoxia | interventions — fluoromisonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 mCi HX4 (Active Comparator): Patient will be injected with [F-18] FMISO
  Interventions: Drug: [F-18] HX4
- 10 mCi FMISO (Active Comparator): Patient will be injected with [F-18] HX4
  Interventions: Drug: [F-18] FMISO

INTERVENTIONS:
Drug: [F-18] FMISO — 10 mCi [F18] HX4 and 10 mCi [F-18] FMISO within 7 days of each other regardless of sequence
  Arms: 10 mCi FMISO
Drug: [F-18] HX4 — 10 mCi [F18] HX4 and 10 mCi [F-18] FMISO within 7 days of each other regardless of sequence
  Arms: 10 mCi HX4

SUMMARY:
Positron Emission Tomography (PET) with fluorine-18 fluoromisonidazole (FMISO) has been used for several years as a non invasive imaging technique to study tumor hypoxia. Several experimental and clinical studies have indicated that FMISO uptake of tissues is correlated with tissue oxygen tension and that FMSO PET allows non-invasive differentiation between hypoxic and normoxic tumors. Currently, FMISO-PET represents the best characterized and validated noninvasive hypoxia imaging technique. Nevertheless, clinical studies have also shown the limitations of FMISO PET. Accumulation of FMISO in hypoxic tumors is relatively low, resulting in a low contrast between hypoxic tumors and surrounding normal tissues. In addition, imaging needs to be started relatively late after tracer injection (about 3 hours post-injection), when a significant percentage of the fluorine-18 label has already decayed and the count statistics of the PET images are relatively low. Because of these limitations, FMISO PET is still only used at a few research centers, despite high clinical interest in hypoxia imaging.

DETAILED DESCRIPTION:
Objective of the study

The aim of this study is to:

* evaluate a hypoxia imaging agent, HX4, in patients with solitary tumors (i.e., locally advanced head and neck cancer)
* gain information on bio-distribution of [F-18]HX4
* compare the PET images of [F-18] FMISO to [F-18]HX4 for resolution, signal to background ratio, and tumor/blood ratio

ELIGIBILITY:
Inclusion Criteria:

* Patient may be male or female and of any race / ethnicity
* Patient is > 18 years old at the time of investigational product administration
* Patient or patient's legally acceptable representative provides written informed consent
* Patient is capable of complying with study procedures
* Patient is capable of communicating with study personnel
* Patient must have histologically confirmed stage III, or IV squamous cell carcinoma of the head and neck whose primary origin was from the oral cavity, oropharynx, hypopharynx, or larynx.
* According to the Karnofsky Performance Status Scale, the patient has a value of ≥ 60% at time of screening
* Patient must have normal organ and renal function as defined:

  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 x institutional upper limits of normal
  * creatinine within normal institutional limits
  * BUN within normal institutional limits
  * PT and PTT < 2.0 x institutional upper limits of normal

Exclusion Criteria:

* Patient is younger than 18 years old at the time of investigational product administration
* Female patient is pregnant or has a positive serum pregnancy test
* Patient is unable to remain still for duration of imaging procedure
* Patient has a history of significant renal disease
* Patient has previously received [F-18]HX4 at any time, or any other investigational product in the past thirty days.
* Patient has been involved in an investigative, radioactive research procedure within the past year
* Inadequate tumor sites or volume to allow for biopsy
* Patient has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete and good quality data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of a hypoxia imaging agent, HX4, in patients with solitary tumors (i.e., locally advanced head and neck cancer) | 6 months

SECONDARY OUTCOMES:
Resolution, signal to background ratio, and tumor/blood ratio of PET images with [F-18] FMISO and [F-18]HX4 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi Hui Guan, MD, Principal Investigator — PET Center, Huashan Hospital, Fudan University
Locations (1):
- PET Center, Huashan Hospital, Fudan University, Shanghai, China